CLINICAL TRIAL: NCT05599776
Title: The Effect of Smart Ring Assisted Physiotherapeutic Intervention on the Risk of Poor Outcome 12 Months After a Total Knee Replacement: a Randomized Controlled Trial
Brief Title: The Effect of Smart Ring Assisted Physiotherapeutic Intervention After TKR
Acronym: SmarTKRing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coxa, Hospital for Joint Replacement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R22078
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Osteo Arthritis Knee
Keywords: total knee replacement; wearable activity tracker; smart ring; physiotherapy

STUDY DESIGN:
Intervention Model Description: The study design is a 2 arm, 1:1 randomized, controlled, single-center trial adhering to Standard Protocol Items: Recommendation for Interventional Trials (SPIRIT) guidelines. The study will be carried out at Coxa Hospital for Joint Replacement (Tampere, Finland), a university-affiliated publicly funded orthopaedic hospital specializing in joint replacement surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group of this trial will receive standard postoperative care which includes physiotherapy appointments 4 weeks and 3 months after the surgery. The 4-week physiotherapy appointment will be at local health center, occupational health clinic or in private physiotherapy clinic and patients are instructed to book the appointments independently according to the standard of care in Coxa Hospital. The 3-month physiotherapy appointment in Coxa Hospital will be carried out by physiotherapists who are dedicated to research projects at Coxa outpatient clinic.
- Intervention group (Experimental): The patients in the intervention group will receive standard physiotherapy care but patients also use smart rings (Oura ring) 3 months postoperatively. Patients will be remotely monitored to follow their recovery from TKR surgery: the study group physiotherapists will follow the patients' activity and sleep and if necessary, make a contact with patient if there seems to low activity indicating difficulties with recovering from the surgery. If there is a constantly decreasing trends in these parameters or patient improvement plateaus, patient is contacted and their status is evaluated by telephone. Based on the information from this contact, the patients may be asked to visit the physiotherapist at the outpatient clinic to assess the situation, and also anesthetist may be consulted on the pain medication. Data collected with the Oura ring will also be used in physiotherapy appointments as a part of therapeutic treatment and guidance.
  Interventions: Other: Smart ring assisted physiotherapeutic intervention

INTERVENTIONS:
Other: Smart ring assisted physiotherapeutic intervention — the effect of a smart ring (Oura), a wearable activity tracker assisted physiotherapeutic intervention on the risk of poor outcome measured on patient reported post-operative outcome (Oxford Knee Score) 12 months after a primary total knee replacement.
  Arms: Intervention group

SUMMARY:
The goal of this randomized controlled trial is to learn about the effect of a wearable activity tracker assisted physiotherapeutic intervention on the risk of poor patient reported outcome after a primary total knee replacement.

The main question it aims to answer is whether a wearable activity tracker assisted physiotherapeutic intervention and remote monitoring may help to decrease the number of the poor patient reported post-operative outcome 12 months after a primary total knee replacement.

Participants will receive standard postoperative care which includes physiotherapy appointments 4 weeks and 3 months after the surgery and they will use smart rings (Oura ring) 3 months postoperatively. Patients will be remotely monitored to follow their recovery from total knee replacement surgery: the study group physiotherapists will follow the patients' activity and sleep and if necessary, make a contact with patient if there seems to low activity indicating difficulties with recovering from the surgery.

Researchers will compare the intervention group to a group of participants who will receive only standard postoperative care with physiotherapy appointments 4 weeks and 3 months, to see if the use of the Oura ring may decrease the number of participants with poor patient reported post-operative outcome after total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary TKA for primary osteoarthritis.
* Patients able to consent and willing to comply with the study protocol.
* Patients aged 18 to 70 years
* Patients is able to use a smartphone and a smart ring.

Exclusion Criteria:

* Patients unwilling to provide informed consent
* >15 degrees varus or valgus, or > 15 degrees fixed flexion deformity
* Physical, emotional, or neurological conditions that would compromise the patient, e.g., poor compliance with postoperative rehabilitation and follow-up (e.g., drug or alcohol abuse, serious mental illness, general neurological conditions, such as Parkinson, MS, etc.)
* Patients unable to attend the study physiotherapy appointments at the outpatient clinic.
* Patients unable to wear Oura ring (example in case of OA or rheumatoid arthritis in the finger joints).
* Patients with cardiac arrhythmia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with poor postoperative outcome | 12 months after total knee replacement surgery

SECONDARY OUTCOMES:
homogeneity of variance in the Oxford Knee Score | 12 months after the surgery
Oxford Knee Score | 3 months after the surgery
  difference between groups
Oxford Knee Score | 6 months after the surgery
  difference between groups
Oxford Knee Score | 12 months after the surgery
  difference between groups
EQ-5D-5L | 3 months after the surgery
  difference in quality of life
EQ-5D-5L | 6 months after the surgery
  difference in quality of life
EQ-5D-5L | 12 months after the surgery
  difference in quality of life
Forgotten Joint Score 12 (FJS-12) | 3 months after the surgery
Forgotten Joint Score 12 (FJS-12) | 6 months after the surgery
Forgotten Joint Score 12 (FJS-12) | 12 months after the surgery
pain at rest using the visual analoque (VAS scale) | 3 months after surgery
pain at rest using the visual analoque (VAS scale) | 6 months after surgery
pain at rest using the visual analoque (VAS scale) | 12 months after surgery
pain while walking using the visual analoque (VAS scale) | 3 months after surgery
pain while walking using the visual analoque (VAS scale) | 6 months after surgery
pain while walking using the visual analoque (VAS scale) | 12 months after surgery
active knee range of motion | 3 months after surgery
active knee range of motion | 12 months after surgery
passive knee range of motion | 3 months after surgery
passive knee range of motion | 12 months after surgery
The patient satisfaction VAS | 12 months after surgery
patient accepted symptom state questions | 12 months after surgery

OTHER OUTCOMES:
the visits to the emergency department | during the 12-month follow-up after surgery
the readmissions to Coxa Hospital | during the 12-month follow-up after surgery
The rate of manipulation under anesthesia | during the 12-month follow-up after surgery
complications | during the 12-month follow-up after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aleksi Reito, MD, PhD, Principal Investigator — Coxa, Hospital for Joint Replacement
Locations (1):
- Coxa Hospital for Joint Replacement, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided
We will share IPD against well-planned research protocol.

REFERENCES:
- [Derived] Hautala J, Koriseva L, Reito A, Mattila V, Eskelinen A. Effect of a smart ring-assisted physiotherapeutic intervention on the postoperative outcomes 12 months after a total knee replacement (SmarTKRing): protocol for a randomised controlled trial. BMJ Open. 2025 May 15;15(5):e091956. doi: 10.1136/bmjopen-2024-091956. PMID 40379331